CLINICAL TRIAL: NCT01880437
Title: A PHASE IB/II STUDY TO EVALUATE THE SAFETY AND EFFICACY OF VISMODEGIB IN RELAPSED/REFRACTORY ACUTE MYELOGENOUS LEUKEMIA (AML) AND RELAPSED/REFRACTORY HIGH-RISK MYELODYSPLASTIC SYNDROME (MDS)
Brief Title: A Study of Vismodegib in Patients With Relapsed/Refractory Acute Myelogenous Leukemia and Relapsed Refractory High-Risk Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GO28852; 2013-001570-14 (EudraCT Number)
Record Dates: First submitted 2013-06-11; First posted 2013-06-19 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndromes, Myelogenous Leukemia, Acute
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid | interventions — Cytarabine; HhAntag691

ARMS (1):
- Vismodegib (Experimental)
  Interventions: Drug: cytarabine; Drug: vismodegib

INTERVENTIONS:
Drug: cytarabine — Cohort 2: 20 mg sc daily for 10 days starting Day 1, with a possible further cycle of 20 mg sc daily for 5 days starting no earlier than Day 29
Drug: vismodegib — Cohorts 1 and 2: 150 mg orally daily
  Other Names: RO5450815

SUMMARY:
This study will assess the safety and efficacy of vismodegib in patients with relapsed/refractory acute myelogenous leukemia (AML) and relapsed/refractory high-risk myelodysplastic syndrome (MDS). Patients in Cohort 1 will receive single-agent vismodegib 150 mg orally daily. In Cohort 2, patients will receive vismodegib 150 mg orally daily in combination with cytarabine 20 mg subcutaneously for 10 days.

Anticipated time on study treatment is until disease progression, intolerable toxicity, or patient withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with documented relapsed or refractory AML, except acute promyelocytic leukemia (APL [M3 subtype]), or relapsed or refractory high-risk MDS (high-risk MDS defined as International Prognostic Scoring System (IPSS) Int-2 or high and >/= 10% blasts in bone marrow)
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Negative serum pregnancy test for women of childbearing potential and use of two forms of contraception while enrolled in the study and for 7 months after the patient discontinues from study
* Male patients with female partners of childbearing potential must agree to use a latex condom and to advise their female partner to use an additional method of contraception during the study and for 2 months after the last dose of vismodegib
* All non-hematological adverse events of any prior chemotherapy, surgery, or radiotherapy must have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade </= 2 prior to starting therapy
* Adequate hepatic and renal function

Exclusion Criteria:

* Prior treatment with a Hh pathway inhibitor
* Prior therapy for the treatment of malignancy within 14 days of Day 1, with the exception of:

Hydroxyurea in patients who need to continue this agent to maintain white blood cell (WBC) counts </= 50,000/mL. Hydroxyurea must be discontinued by Day 14 of the study

* Current evidence of active central nervous system (CNS) leukemia
* Any other active malignancy (except non-melanoma skin cancer or carcinoma in situ of the cervix)
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

Unstable angina, symptomatic or otherwise uncontrolled arrhythmia requiring medication (does not include stable, lone atrial fibrillation), or myocardial infarction </= 6 months before study treatment start Any active (acute or chronic) or uncontrolled infection/disorders that impair the ability to evaluate the patient or for the patient to complete the study

* Pregnant or breast-feeding women
* Patients who refuse to potentially receive blood products and/or have a severe hypersensitivity to blood products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- United States (5):
  - Stanford, California
  - Ann Arbor, Michigan
  - Kansas City, Missouri
  - New York, New York
  - Houston, Texas
- Canada (3):
  - Edmonton, Alberta
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (5):
  - Braunschweig
  - Essen
  - Hamburg
  - Heidelberg
  - Münster

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 47 participants were screened; of which,7 participants failed screening and 2 participants were erroneously entered but did not receive study drug.A total of 38 participants were enrolled and treated. It was planned to enroll 2 cohorts; Cohort 1 (vismodegib) and Cohort 2 (vismodegib + cytarabine).
Pre-assignment Details: Based on lower-than-expected efficacy observed in interim data review, study was terminated prior to initiation of Cohort 2. Results are reported as per subgroups of Cohort 1: "Poor Risk Cytogenetics", "FLT-3 Mutation Positive", "Neither Poor Risk Cytogenetics Nor FLT-3", unless otherwise specified.
Groups:
- Poor Risk Cytogenetics: Participants with relapsed/refractory acute myeloid leukemia (AML) or relapsed/refractory high-risk myelodysplastic syndrome (MDS) falling under 'poor risk cytogenetics' subgroup received oral 150 milligrams (mg) dose of vismodegib capsule once daily until disease progression, intolerable toxicity most probably attributable to vismodegib, or participant withdrawal of consent.
- FLT-3 Mutation Positive: Participants with relapsed/refractory AML or relapsed/refractory high-risk MDS falling under 'FLT-3 mutation positive' subgroup received oral 150 mg dose of vismodegib capsule once daily until disease progression, intolerable toxicity most probably attributable to vismodegib, or participant withdrawal of consent.
- Neither Poor Risk Cytogenetics Nor FLT-3: Participants with relapsed/refractory AML or relapsed/refractory high-risk MDS falling neither under 'poor risk cytogenetics' nor 'FLT-3 mutation positive' subgroup were included in this group and received oral 150 mg dose of vismodegib capsule once daily until disease progression, intolerable toxicity most probably attributable to vismodegib, or participant withdrawal of consent.
Period: Overall Study
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT-3
Started | 15 | 4 | 19
Completed | 0 | 0 | 0
Not Completed | 15 | 4 | 19
Not completed — Death | 12 | 4 | 17
Not completed — Study terminated by Sponsor | 3 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Poor Risk Cytogenetics: Participants with relapsed/refractory AML or relapsed/refractory high-risk MDS falling under 'poor risk cytogenetics' subgroup received oral 150 mg dose of vismodegib capsule once daily until disease progression, intolerable toxicity most probably attributable to vismodegib, or participant withdrawal of consent.
- Total: Total of all reporting groups
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT-3 | Total
Number analyzed (Participants) | 15 | 4 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (20.7) | 54.5 (5.9) | 66.2 (14.7) | 63.1 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 9 | 17
  Male | 9 | 2 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response (CR) or CR With Incomplete Blood Count Recovery (CRi) or Morphologic Leukemia Free State (MLFS) or Partial Response (PR) at Week 8
Description: CR was defined as achieved if the neutrophils count was greater than (>) 1000 cells per microliter (µL), platelets count >100000/µL, bone marrow blasts percentage (%) less than (<) 5, no Auer rods (clumps of azurophilic granular material that form elongated needles seen in the cytoplasm of leukemic blasts), no transfusion requirements and no signs of extra medullary disease (EMD). CRi was defined if either of the cell (neutrophil or platelet) lineage was not recovered (neutrophils >1000 cells/µL or Not applicable [NA] or platelets count >100000/µL or NA), bone marrow blasts <5% with no Auer rods and confirmed by flow cytometry with no signs of EMD. MLFS (neutrophil and platelet criteria were NA) was defined as bone marrow blasts <5% with no Auer rods and confirmed by flow cytometry with no signs of EMD. PR was defined as neutrophils count >1000 cells/µL, platelets count >100000/µL, and >50% decrease from baseline to a range of 5-25% of bone marrow blasts or blasts <5% with Auer rods.
Time Frame: Week 8
Population: As the primary efficacy time-point (Week 8) was not reached for all participants due to study termination based on interim data analysis, the analysis of this outcome measure could not be performed, as per planned analysis.
Groups:
- Neither Poor Risk Cytogenetics Nor FLT3: Participants with relapsed/refractory AML or relapsed/refractory high-risk MDS falling neither under 'poor risk cytogenetics' nor 'FLT-3 mutation positive' subgroup were included in this group and received oral 150 mg dose of vismodegib capsule once daily until disease progression, intolerable toxicity most probably attributable to vismodegib, or participant withdrawal of consent.
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants With CR, CRi, MLFS or PR at Anytime During Study Treatment
Description: CR was defined as achieved if the neutrophils count >1000 cells/µL, platelets count >100000/µL, bone marrow blasts <5%, no Auer rods (clumps of azurophilic granular material that form elongated needles seen in the cytoplasm of leukemic blasts), no transfusion requirements and no signs of EMD. CRi was defined if either of the cell (neutrophil or platelet) lineage was not recovered (neutrophils > 1000 cells/µL or NA or platelets count >100000/µL or NA, bone marrow blasts <5% with no Auer rods and confirmed by flow cytometry with no signs of EMD. MLFS (neutrophil and platelet criteria were NA) was defined as bone marrow blasts <5% with no Auer rods and confirmed by flow cytometry with no signs of EMD. PR was defined as neutrophils count >1000 cells/µL, platelets count >100000/µL, and >50% decrease from baseline to a range of 5-25% of bone marrow blasts or blasts <5% with Auer rods. The 95% confidence intervals (CI) were constructed using Blyth-Still-Cassella method.
Time Frame: Up to 30 days of last dose of study drug (maximum treatment duration = 225 days)
Population: Efficacy analysis population included all enrolled participants. Here "number of participants analyzed" included participants who were evaluable for tumor response at anytime during the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT3
Number analyzed (Participants) | 13 | 4 | 16
percentage of participants
  CR | 0 [0.00 to 22.51] | 0 [0.00 to 52.71] | 0 [0.00 to 19.75]
  CRi | 0 [0.00 to 22.51] | 0 [0.00 to 52.71] | 6.3 [0.32 to 29.88]
  MLFS | 0 [0.00 to 22.51] | 0 [0.00 to 52.71] | 0 [0.00 to 19.75]
  PR | 0 [0.00 to 22.51] | 0 [0.00 to 52.71] | 6.3 [0.32 to 29.88]

3. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR is defined as the time from the first occurrence of a documented overall response to the time of relapse, as determined by the investigator using International Working Group (IWG) criteria (Participants not falling under any of the response criteria [CR or CRi or MLFS or PR] described under outcome measure 1 were considered as non-responders) or death from any cause during the study (defined as death within 30 days after the last dose of study drug).
Time Frame: Up to 30 days of last dose of study drug (maximum treatment duration = 225 days)
Population: Efficacy population including participants who were considered as responders.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT3
Number analyzed (Participants) | 0 | 0 | 2
weeks
  DOR of participants with CRi (n=0,0,1) |  |  | 13 [NA to NA] — The 95% CI was not estimable as only 1 participant was evaluable.
  DOR of participants with PR (n=0,0,1) |  |  | 6.1 [NA to NA] — The 95% CI was not estimable as only 1 participant was evaluable.

4. Secondary Outcome: Median Overall Survival (OS) Time
Description: OS was defined as the time from start of study drug to death from any cause. OS was estimated using Kaplan-Meier analysis. Participants alive at the last date known to be alive were censored for the analysis.
Time Frame: Up to death or 30 days of last dose of study drug (maximum treatment duration = 225 days)
Population: Efficacy analysis population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT-3
Number analyzed (Participants) | 15 | 4 | 19
months | 3.38 [2.37 to 4.83] | 1.43 [0.33 to 3.94] | 3.65 [1.94 to 5.36]

5. Secondary Outcome: Percentage of Participants With an Event of Death During the Study
Time Frame: Up to death or 30 days of last dose of study drug (maximum treatment duration = 225 days)
Population: Efficacy analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT-3
Number analyzed (Participants) | 15 | 4 | 19
percentage of participants | 80.0 | 100.0 | 89.5

6. Secondary Outcome: Pharmacokinetics (PK): Steady-state Plasma Concentration of Vismodegib
Description: PK data was planned to be reported only if the results of Cohort 2 are available.
Time Frame: Predose on Days 8, 29 and 57
Population: As the study was terminated prior to Cohort 2 enrollment, PK analysis could not be performed, as planned.
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT-3
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Area Under the Concentration-time Curve (AUC) of Cytarabine
Description: PK data was planned to be reported only if the results of Cohort 2 are available.
Time Frame: Predose, 0.25, 0.5, 1, 3, 6 hours post-dose on Days 1, 8 and 29
Population: No participants were enrolled as the study was terminated prior to the initiation of Cohort 2.
Groups:
- Planned Cohort 2: Participants in Cohort 2 were planned to receive low-dose subcutaneous injections of cytarabine in combination with continuous daily vismodegib (150 mg orally).
Arm/Group | Planned Cohort 2
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From screening until study completion or early termination visit (Up to 14 months)
Arm/Group | Poor Risk Cytogenetics | FLT-3 Mutation Positive | Neither Poor Risk Cytogenetics Nor FLT-3
Serious Adverse Events (participants affected / at risk) | 10/15 | 3/4 | 13/19
Other Adverse Events (participants affected / at risk) | 13/15 | 4/4 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poor Risk Cytogenetics (N=15) | FLT-3 Mutation Positive (N=4) | Neither Poor Risk Cytogenetics Nor FLT-3 (N=19)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 6
Graft versus host disease (Immune system disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 3 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 3
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Vaginal abscess (Infections and infestations) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Central venous catheterisation (Surgical and medical procedures) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Poor Risk Cytogenetics (N=15) | FLT-3 Mutation Positive (N=4) | Neither Poor Risk Cytogenetics Nor FLT-3 (N=19)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 2
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Scleral discolouration (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 4 | 0 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 0 | 10
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4
Asthenia (General disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 1 | 2
Early satiety (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 2 | 5
Feeling cold (General disorders) | 0 | 0 | 1
Localised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 4 | 0 | 4
Pain (General disorders) | 1 | 0 | 3
Peripheral swelling (General disorders) | 2 | 0 | 1
Pyrexia (General disorders) | 3 | 3 | 5
Candida infection (Infections and infestations) | 0 | 0 | 1
Catheter site infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 2
Erysipelas (Infections and infestations) | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 2
Liver abscess (Infections and infestations) | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 2
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 2
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 1
Cardiac murmur (Investigations) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2
Platelet count decreased (Investigations) | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 6
Dysgeusia (Nervous system disorders) | 4 | 1 | 7
Headache (Nervous system disorders) | 2 | 1 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1
Orthostatic intolerance (Nervous system disorders) | 0 | 0 | 1
Radicular pain (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2
Disorientation (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Vulval ulceration (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pain (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 3
Hypertension (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 4
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0
Vasculitis (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This study was prematurely terminated because of lower-than-expected efficacy observed in interim data analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.